CLINICAL TRIAL: NCT01788501
Title: Tacrolimus/Methotrexate Versus Cyclosporine/Methotrexate for Prophylaxis of Graft Versus Host Disease in Paediatric Patients
Brief Title: Tacrolimus/Methotrexate Versus Cyclosporine/Methotrexate for Prophylaxis of Graft Versus Host Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyoung Jin Kang, professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SNUCP_001
Record Dates: First submitted 2012-11-25; First posted 2013-02-11 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Tacrolimus; Cyclosporine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacrolimus/Methotrexate (Experimental): Tacrolimus D-1~D20: iv infusion, q24hr (first daily dose: 0.03mg/kg) D20~D100: po q12hr (first daily dose: the quadruple of last iv dose) Dose modification according to therapeutic drug monitoring(TDM) (10-20ng/ml)
  Methotrexate D1: 15mg/m2 iv push D3,6,(11): 10mg/m2 iv push
  Interventions: Drug: Tacrolimus; Drug: Methotrexate
- Cyclosporine/Methotrexate (Active Comparator): Cyclosporine D-1~D20: iv infusion, q24hr (first daily dose: 3mg/kg) D20~D100: po q12hr (first daily dose: the 3 times of last iv dose) Dose modification according to TDM (200-300ng/ml)
  Methotrexate D1: 15mg/m2 iv push D3,6,(11): 10mg/m2 iv push
  Interventions: Drug: Cyclosporine; Drug: Methotrexate

INTERVENTIONS:
Drug: Tacrolimus — D-1~D20: iv infusion, q24hr (first daily dose: 0.03mg/kg) D20~D100: po q12hr (first daily dose: the quadruple of last iv dose) Dose modification according to TDM (10-20ng/ml)
  Arms: Tacrolimus/Methotrexate
Drug: Cyclosporine — D-1~D20: iv infusion, q24hr (first daily dose: 3mg/kg) D20~D100: po q12hr (first daily dose: the 3 times of last iv dose) Dose modification according to TDM (200-300ng/ml)
  Arms: Cyclosporine/Methotrexate
Drug: Methotrexate — D1: 15mg/m2 iv push D3,6,(11): 10mg/m2 iv push

SUMMARY:
This study aims to compare efficacy and safety of tacrolimus/methotrexate with cyclosporine/methotrexate for graft versus host disease prophylaxis in paediatric allogeneic hematopoietic stem cell transplantation patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hematological malignancy
* Age under 18 years old
* Serum bilirubin less than 1.5 X upper limit of normal
* Aspartate transaminase, Alanine transaminase less than 2.5 X upper limit of normal
* Alkaline phosphatase less than 2.5 X upper limit of normal
* Serum creatinine less than 1.5 X upper limit of normal
* Agrees to participate, and informed consent signed

Exclusion Criteria:

* Evidence of HIV infection
* Documented uncontrolled disease (infections)
* Prior transplantation (hematopoietic stem cell or solid organs)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
incidence of grade II-IV acute graft versus host disease | day 100 post transplantation
  Overall grade I graft-versus-host disease denoted stage 1 to 2 skin involvement with no liver or gut involvement. Overall grade II graft-versus-host disease denoted stage 3 skin involvement or stage 1 liver or gut involvement. Overall grade III graft-versus-host disease denoted stage 4 skin involvement or stage 2 to 4 liver or gut involvement without graft-versus-host disease as a major contributing cause of death. And Overall grade IV graft-versus-host disease denoted stage 4 skin involvement or stage 2 to 4 liver or gut involvement with graft-versus-host disease as a major contributing cause of death.

SECONDARY OUTCOMES:
incidence of infection | day 100 post transplantation
  Fever would be categorized as fever occured before engraftment and after engraftment. If microbiologically documented, pathogen would be specified.
incidence of adverse drug reactions | day 100 post transplantation
  adverse drug reactions would be measured by Common Terminology Criteria for Adverse Events v3. And for determinating the likelihood of whether an adverse drug reaction is actually due to the drug, Naranjo algorithm would be used

CONTACTS AND LOCATIONS:
Overall Officials: JungMi Oh, Pharm.D, Principal Investigator — Seoul National University College of Pharmacy
Locations (3):
- South Korea (3):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No